CLINICAL TRIAL: NCT06712433
Title: Bacterial Decolonization Plus Intraoperative Indocyanine Green Angiography for Soft Tissue Sarcomas of the Lower Extremity Receiving Preoperative Radiotherapy (CONCERTO)
Brief Title: Bacterial Decolonization Plus Intraoperative Angiography for Soft Tissue Sarcomas Receiving Preoperative Radiotherapy (CONCERTO)
Acronym: CONCERTO
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Adam Olson (Other)
Collaborators: Pittsburgh Cure Sarcoma (Unknown)
Responsible Party: Sponsor-Investigator, Adam Olson, Assistant Professor, Radiation Oncology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 24-080
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Sarcoma,Soft Tissue
Keywords: bacterial decolonization (BD); external beam radiotherapy (RT); wide local excision (WLE); intraoperative IICG angiography
MeSH Terms: conditions — Sarcoma | interventions — chlorhexidine gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BD + Intranasal Mupirocin + Chlorhexidine (Experimental): Bacterial Decolonization with 2% intranasal mupirocin ointment twice daily (BID) and 4% chlorhexidine gluconate body cleanser, once daily (QD) for 5 consecutive days prior to RT, and this will be repeated for 5 days every 2 weeks throughout Radiation Therapy.
  The treatment will also be administered for 5 consecutive days prior to index surgery. RT can be prescribed in one of three dose/fractionation regimens at the investigator's discretion: 50 Gy in 25 fractions, 42.75 Gy in 15 fractions, or 36 Gy in 18 fractions
  Interventions: Drug: 2% intranasal mupirocin ointment; Drug: 4% chlorhexidine gluconate body cleanser

INTERVENTIONS:
Drug: 2% intranasal mupirocin ointment — Mupirocin nasal ointment is used to treat or prevent infections in the nose due to certain strains of Staphylococcus aureus bacteria. This medicine works by killing bacteria or preventing their growth.
Drug: 4% chlorhexidine gluconate body cleanser — Chlorhexidine Gluconate (CHG) Solution Antiseptic Skin Cleanser solution is a topical skin cleanser that keeps working after it is used. CHG is a strong antiseptic (liquid used to kill germs and bacteria) that lowers the risk of infection.
  Other Names: Hibiclens®

SUMMARY:
This trial will investigate the combination of two low-cost, non-toxic strategies to assess whether they can reduce the risk of acute major wound complications in soft tissue sarcoma of the lower extremity. Intranasal mupirocin ointment twice daily and chlorhexidine body cleanser once daily for 5 days prior to radiation therapy and repeated for 5 days every 2 weeks during radiation therapy may significantly reduce the risk of acute radiation dermatitis. That, along with use of indocyanine green (ICG) angiography at the time of wound closure.

DETAILED DESCRIPTION:
Strategies to reduce the risk of acute wound complications have historically been mostly unsuccessful. In soft tissue sarcomas, a prior study showed that the use of indocyanine green (ICG) angiography at the time of wound closure was associated with a reduction in wound dehiscence and infection when compared to historical controls. Cutaneous colonization of S. aureus has been implicated in severe cases of radiation dermatitis. Some known risk factors for acute major wound complications for patients with sarcomas are anatomic location in the lower extremity, preoperative radiation therapy, larger tumors, comorbidities (e.g., diabetes mellitus, tobacco usage, vascular disease, and obesity), tumors <3mm from skin surface, and the development of grade ≥ 2 acute radiation dermatitis. Both large tumors and lower extremity location can increase the likelihood of seroma formation, which can act as a nidus for infection and subsequent wound complication. Rationale for this trial includes prior studies of treating patients with a bacterial decolonization (BD) protocol of intranasal mupirocin ointment twice daily and chlorhexidine body cleanser once daily for 5 days prior to RT and repeated for 5 days every 2 weeks during radiation therapy that show significantly reduced risk of acute radiation dermatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
2. Newly diagnosed soft tissue sarcoma arising from the lower extremity (defined as the tumor center arising at the level of the iliac crest or below)
3. Eligible for wide local excision
4. Eligible for external beam radiation therapy
5. Negative serum pregnancy test for women of childbearing potential < 28 days prior to RT.
6. Informed consent signed and dated to participate in the study.
7. Willingness and ability to comply

Exclusion Criteria:

1. Allergy to mupirocin and/or chlorhexidine
2. Active dermatologic condition in RT field
3. Tumor size > 32cm
4. Prior RT overlapping with fields
5. Concurrent/prior invasive malignancy that could potentially interfere with proposed treatment. Individual cases can be discussed with PI prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2026-09-30 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and type of acute major wound complications | Up to 24 months
  Incidence and type of acute major wound complications: One or more of the following events occurring within 4 months of index sarcoma surgery including: 1). A secondary operation under general or regional anesthesia for wound repair (debridement, operative drainage, and secondary wound closure including rotationplasty, free flaps, or skin grafts), 2). Wound management without secondary operation, such, An invasive procedure without general or regional anesthesia (such as aspiration of seroma), Readmission for wound care such as intravenous antibiotics, or Persistent deep packing for 120 days or longer.

SECONDARY OUTCOMES:
1-year Local control | At 1 year
  Local control is defined as the proportion of patients without clinical evidence of local recurrence. This will be reported as will a cumulative incidence curve of local failures, considering using death as a competing risk, using the cumulative incidence function method.
2-year Local control | At 2 years
  Local control is defined as the proportion of patients without clinical evidence of local recurrence. This will be reported as will a cumulative incidence curve of local failures, considering using death as a competing risk, using the cumulative incidence function method.
Progression-free survival (PFS) | Up to 24 months
  Median number of months from start of treatment until the date of disease progression or death from any cause.
Overall survival (OS) | Up to 24 months
  Median number of months from start of treatment until death from any cause.
Musculoskeletal Tumour Society Score [MSTS] | Up to 24 months
  The MSTS is a patient questionnaire for assessing physical function after medical treatment, surgery, and physiotherapy in patients with malignant bone tumors in specific extremities. The MSTS questionnaire consists of six domains, each scored on a scale from 0 to 5, with a higher score indicating better function. The total score, ranging from 0 (maximum disability) to 30 (no impairment), can be transformed to a point scale of 0 to 100.
Toronto Extremity Salvage Score [TESS] | Up to 24 months
  TESS represents the gold standard for assessing function after surgery for muscle and bone tumors, as it has been tested for validity and reliability, and extremity-specifically defines disability, handicap, change in physical function depending on the therapeutic intervention and the patient's need for an aid. The TESS questionnaire has both upper and lower extremity versions. Twenty-nine items are rated on a scale from one to five, with five representing normal activity. The result ranges from 0 to 100, with 100 being the best score.
Adverse Events and Serious Adverse Events related to intervention(s) | Up to 24 months
  Adverse Events and Serious Adverse Events per CTCAE v5.0 that attributed to study intervention(s).
Frequency of late toxicities | Up to 24 months
  Acute toxicities are defined as toxicity occurring during preoperative RT, after RT and prior to surgery, and within 90 days of index resection, assessed using CTCAE v5.0.
Change in type of actual surgical closures | At surgery
  Tabulation of the initial surgical closure intended, and the actual surgical closure used at the time of index resection. Descriptive statistics will be used to summarize these assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Adam M Olson, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Centers, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No